CLINICAL TRIAL: NCT04742790
Title: Clinical Calibration and Evaluation of the QSPainRelief Platform in Patients With Disabling Pain Using Functional Biomarkers of Nociception, Sedation and Cognition
Brief Title: QSPainRelief-patientCNS : Clinical Biomarkers of Nociception, Sedation and Cognition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: QSPainRelief-patientCNS; VER.01-30.06.2020 (Other: Comité d'Ethique Hospitalo-Facultaire de l'UCLouvain)
Record Dates: First submitted 2021-01-26; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Post-operative Pain
Keywords: acute pain; persistent pain; sedation
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Laser-Evoked Potentials; Patient Reported Outcome Measures

STUDY DESIGN:
Intervention Model Description: Monocentric prospective longitudinal study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): The study will recruit volunteers (1) suffering from disabling post-operative pain for more than two weeks following surgery (thoracotomy, sternotomy and breast cancer surgery), (2) currently being treated for their post-operative pain with an opioid analgesic - along with possible other treatments - and (3) for which the treating physician is about to introduce an additional non-opioid drug for the treatment of their pain (e.g. an antiepileptic or an anti-depressant).
  Interventions: Diagnostic Test: Scalp electroencephalography (EEG); Diagnostic Test: Laser-evoked potentials (LEPs); Diagnostic Test: Cognitive auditory-evoked potentials (P300); Diagnostic Test: Cervical somatosensory-evoked potentials; Diagnostic Test: Pupillometry; Diagnostic Test: Saccadic Peak Velocity; Diagnostic Test: Adaptive tracking test; Diagnostic Test: Body Sway Test; Diagnostic Test: N-back working memory test; Other: Patient-reported outcomes

INTERVENTIONS:
Diagnostic Test: Scalp electroencephalography (EEG) — Resting EEG will be recorded before initiation of the combination treatment (visit 1) and 7-10 days after treatment (visit 2). Drug-induced sedation-related changes in the EEG frequency spectrum. Five minutes of resting EEG eyes-open will be recorded in a quiet room while participants are asked to focus on an image displayed on a wall. Then, they will be asked to close their eyes for an additional 2 minutes. The alpha power ratio eyes open/eyes closed will be computed (alpha attenuation coefficient; Kaida et al., 2006). Changes in this coefficient will be used as a measure of drug-induced sedation.
  Other Names: Biomarker of sedation
Diagnostic Test: Laser-evoked potentials (LEPs) — Laser-evoked potentials (LEPs) will be recorded before (visit 1) and 7-10 after (visit 2) initiating the combination treatment. Short pulses (50-100 ms) of radiant heat generated by a C02 laser stimulator will be applied to the skin of the left or right hand dorm to briefly and selectively activate heat-sensitive pain receptors. A concomitant EEG recordings will be used to measure the amplitude and latency of the elicited laser-evoked potentials. Changes in LEP amplitude (expressed as percentage of change) will be used as a measure of drug-induced effects on the state of the thermonociceptive system.
  Other Names: Biomarker of nociception (brain)
Diagnostic Test: Cognitive auditory-evoked potentials (P300) — Cognitive auditory-evoked potentials will be recorded before (visit 1) and 7-10 after (visit 2) initiating the combination treatment. Short-lasting auditory tones will be delivered using a three-stimulus oddball paradigm combining standard tones (90% of stimuli), slightly different target tones that the subject must attend and detect (10% of stimuli), and strongly different distractor non-target tones (10% of stimuli). The stimuli will be delivered binaurally using headphones. Participants will be instructed to press a button when they detect a target tone, and to ignore the standard and distractor non-target tones. The EEG recordings will be used to measure the amplitude and latency of the cognitive P3a and P3b potentials (Komerchero & Polich 1999). Changes in P3a/P3b amplitude will be used as a measure of drug-induced effects on cognition (expressed as percentage of change).
  Other Names: Biomarker of cognition
Diagnostic Test: Cervical somatosensory-evoked potentials — Cervical spinal-cord evoked potentials will be recorded before (visit 1) and 7-10 after (visit 2) initiating the combination treatment. The responses will be elicited by transcutaneous electrical stimulation of the median nerve. The N13 component of this response is mediated by large myelinated non-nociceptive fibers and reflects a segmental postsynaptic response of dorsal horn interneurons at the level of lumbar spinal cord (Cruccu et al., 2008). Changes in magnitude of the N13 will be used as a measure of drug-induced effects on spinal cord function (expressed as percentage of change).
  Other Names: Biomarker of nociception (spinal)
Diagnostic Test: Pupillometry — Pupillometry measurements will be performed before (visit 1) and 7-10 after (visit 2) initiating the combination treatment. Pupillometry has been proposed as a method to assess opioid pharmacodynamics. The extent of pupil dilatation can provide an index of nociceptive input via autonomic innervation of the iris muscles, while the extent of the attenuation of this pupillary response during exposure to opioid analgesics could provide an index of pharmacological effects reflecting the extent of opioid receptor occupancy in the CNS. Pupillometry (static pupil diameter, variability of pupil diameter [variation coefficient of pupillary dilation, VCPD, Charier et al. 2017]), light-evoked speed of pupil constriction [maximum pupil constriction velocity, PCV, Connely et al., 2014]) will be measured using a handheld pupillometry device routinely used for clinical evaluations.
Diagnostic Test: Saccadic Peak Velocity — The saccadic peak velocity (SPV; m/s) will be measured before before (visit 1) and 7-10 after (visit 2) initiating the combination treatment. Saccadic peak velocity is one of the most sensitive parameters for sedation. Recording of eye movements will be performed in a quiet room with dimmed lightning. Average values of saccadic peak velocity (expressed as degrees/second) of all correct saccades will be measured.
Diagnostic Test: Adaptive tracking test — The test will be performed before (visit 1) and 7-10 after (visit 2) initiating the combination treatment. Adaptive tracking is a pursuit-tracking task sensitive to impairment of eye-hand coordination by drugs. It has been proven useful for measuring CNS effects of alcohol, various other psychoactive drugs, and sleep deprivation.
Diagnostic Test: Body Sway Test — Body sway will be assessed before (visit 1) and 7-10 after (visit 2) initiating the combination treatment, using a body sway meter and with eyes closed. The body sway meter allows measurement of body movements in a single plane, providing a measure of postural stability. The method has been used to demonstrate effects of sleep deprivation, ethanol and psychoactive drugs. All body movements over a 2-min period are integrated and expressed as millimeters of sway.
Diagnostic Test: N-back working memory test — Working memory performance will be assessed before (visit 1) and 7-10 after (visit 2) initiating the combination treatment. In this test, a series of letters are shown to the participant on a computer screen. The test includes three conditions with increased working memory load. The "0-back" condition simply requires to indicate whether the presented letter is the letter "X" or another letter. In the "1-back" condition, participants are requested to indicate whether the displayed letter is identical to the preceding letter. In the "2-back" condition, participants are required indicate whether the letter is repeated with one other letter in between (e.g., B … C … B).
Other: Patient-reported outcomes — Before (visit 1) and 7-10 after (visit 2) initiating the combination treatment, but also daily between the two visits, 14 days, 1 month, 3 months and 6 months after treatment initiation, patient-reported outcomes will be collected to assess clinical effects and side-effects of the combination treatmen These include the short form of the Brief Pain Inventory (BPI), the PROMIS PQ-NEURO score for neuropathic pain, the Stanford Sleepiness Scale (SSS), and the PROMIS Neuro-QOL self-assessment of cognitive functioning.

SUMMARY:
QSPainRelief-patientCNS is a monocentric prospective longitudinal study conducted in patients suffering from disabling post-surgical pain for which the treating physician is about to prescribe a given drug combination for the treatment of their pain with the aim of identifying measures of drug-induced effects on CNS activity that could be used as biomarkers of real-life clinical outcome, both in terms of desired treatment effects (treatment-induced pain relief) but also in terms of undesired treatment effects (treatment-induced sedation and treatment-induced cognitive dysfunction).

DETAILED DESCRIPTION:
QSPainRelief-patientCNS is one of three clinical studies that will be conducted as part of the QSPainRelief project funded by the European Union's Horizon 2020 research and innovation program (grant agreement 848068; http://qspainrelief.eu).

Chronic pain is a complex disease affecting about 20% of Europeans, and up to 60% of patients with chronic pain do not experience adequate pain relief from currently available analgesic combinational therapies and/or suffer confounding adverse effects. Of the many conceivable combinations, only a few have been studied in formal clinical trials. Thus, physicians have to rely on clinical experience when treating chronic pain patients. The vision of the QSPainRelief project is that alternative novel drug combinations with improved analgesic and reduced adverse effects can be identified and assessed by mechanism-based Quantitative Systems Pharmacology (QSP) in silico modelling. The QSPainRelief consortium will setup, calibrate and validate an in silico QSPainRelief platform which integrates recently developed (1) physiologically based pharmacokinetic models to quantitate and adequately predict drug pharmacokinetics in human CNS, (2) target-binding kinetic models; (3) cellular signaling models and (4) a proprietary neural circuit model to quantitate the drug effects on the activity of relevant brain neuronal networks, that also adequately predicts clinical outcome.

Calibration of the QSPainRelief platform modelling the biological processes and neuronal circuits underlying the pain relief and adverse effects induced by drug combinations requires patient data on how different drug combinations affect the central processing of nociceptive input, the central processes underlying pain modulation, as well as the central nervous system (CNS) networks underlying drug-induced adverse effects. After calibration of the QSPainRelief platform, additional patient data is required to evaluate the ability of the platform to actually predict CNS effects of drug combinations in patients. Finally, real-world evidence is needed to relate the effects of drug combinations on CNS activity with the therapeutic and adverse effects self-reported by the patients.

The aims of the QSPainRelief-patientCNS study are thus two-fold.

The first aim is to obtain data from a first set of 60 patients to calibrate the QSPainRelief platform, and from a second set of 120 patients to evaluate the ability of the QSPainRelief platform to predict therapeutic and adverse effects of drug combinations. It will focus on pain relief and its impact on daily life activities as therapeutic effects, and on drug-induced sedation, drug-induced cognitive dysfunction (memory and attention) and pain medication misuse as adverse effects. These adverse effects have been chosen because (1) CNS biomarkers sensitive to drug-induced sedation and drug-induced cognitive dysfunction can be readily obtained using non-invasive measurements of the electroencephalogram (EEG) and (2) the chosen adverse effects can be assessed in patients after a short treatment period using validated patient-reported outcome measures (PROMs).

The second aim is to identify measures of drug-induced effects on CNS activity that could be used as biomarkers of real-life clinical outcome, both in terms of desired treatment effects (treatment-induced pain relief) but also in terms of undesired treatment effects (treatment-induced sedation and treatment-induced cognitive dysfunction).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years.
* Presence of disabling post-operative pain for more than two weeks following thoracotomy, sternotomy or breast cancer surgery.
* Current treatment of their post-operative pain with an opioid analgesic (along with possible other drugs).
* Decision by the treating physician to introduce an additional non-opioid treatment for their post-operative pain such as (but not necessarily) an antiepileptic or an anti-depressant.
* Capacity to understand and voluntarily sign an informed consent form.

Exclusion Criteria:

* Insufficient French language skills.
* Planned chemotherapy, hormonotherapy or radiotherapy during the time interval between Visits 1 and 2.
* Clinically evident psychiatric disease that is likely to interfere with the study, according to judgment by the investigator.
* History of peripheral or central nervous system disease before the surgical intervention.
* Dermatological condition involving the sensory testing areas.
* Severe alcohol use disorder (as defined in DSM-5).
* Severe sedative, hypnotic of anxiolytic-related use disorder (as defined in DSM-5).
* Any other mild, moderate or severe substance use disorder except tobacco and caffeine (as defined in DSM-5).
* Consumption of recreational drugs, including cannabis, in the last 4 weeks prior to the study.
* Signs of polyneuropathy at clinical examination.
* Signs of a neurological deficit due to a CNS lesion or dysfunction at clinical examination.
* Any other reason to exclude the subject because it may interfere with the study, according to judgment by the investigator. The reason will be documented.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between change in magnitude of laser-evoked brain potentials (LEP) and change in the Brief Pain Inventory (BPI) pain severity score | three months
  To assess whether inter-individual differences in the drug-induced change in the magnitude of LEPs (in microvolts) predicts pain relief, the post-drug-combination vs. pre-drug-combination change in magnitude of LEPs between Visit 1 and Visit 2 (expressed as percentage of change between the two visits) will be correlated with the post-drug-combination minus pre-drug-combination change in the pain severity score obtained from the BPI (score between 0 and 40; Gjeilo et al., 2007) between Visit 1 and Month 3.
Correlation between change in the alpha attenuation coefficient (AAC) and change in the Stanford Sleepiness Scale (SSS) | 10 days
  To assess whether inter-individual differences in the drug-induced change in AAC (ratio between alpha-band power eyes closed vs. eyes open; Kaida et al., 2006) predicts self-reported sleepiness, the post-drug-combination minus pre-drug combination change in the AAC measured in the resting EEG between Visits 1 and 2 will be correlated with the post-drug-combination minus pre-drug-combination change in self-reported sleepiness assessed using the Stanford Sleepiness Scale (SSS; score between 1 and 7) between Visits 1 and 2.
Correlation between change in magnitude of cognitive P3b potential and change in the PROMIS Neuro-QOL score for cognitive function | 10 days
  To assess whether inter-individual differences in the drug-induced change in magnitude of the P3b component of auditory-evoked potentials (in microvolts; Komerchero & Polich 1999) predicts self-reported cognitive dysfunction, the post-drug-combination vs. pre-drug-combination change in P3b magnitude between Visits 1 and 2 (expressed as percentage of change) will be correlated with the post-drug-combination minus pre-drug-combination change in self-reported cognitive dysfunction assessed using the short-form cognitive function measurement of the PROMIS Neuro-QOL (Quality of Life in Neurological Disorders) between Visits 1 and 2 (standardized T score for "cognitive function", having a mean of 50 and a standard deviation of 10 in a reference population).

SECONDARY OUTCOMES:
Correlation between change in magnitude of the N13 spinal-cord evoked potential and change in the PQ-NEURO score for neuropathic pain | 10 days
  To assess whether inter-individual differences in the drug-induced change in magnitude of the N13 spinal-cord evoked potential (in microvolts; Cruccu et al., 2008) predicts changes in self-reported signs of neuropathic pain, the post-drug-combination vs. pre-drug-combination change in amplitude of the N13 (expressed as percentage of change) between Visits 1 and 2 will be correlated to the post-drug-combination minus pre-drug-combination change in the PROMIS measure of neuropathic pain quality (PQ-NEURO ; Askew et al. 2016) between Visits 1 and 2 (standardized T score with a mean of 50 and standard deviation of 10 in a reference population).
Correlation between change in the variation coefficient of pupillary dilation (VCPD) and change in the Brief Pain Inventory (BPI) score | 10 days
  To assess whether inter-individual differences in the drug-induced change in the VCPD (Charier et al., 2017) predicts pain relief, the post-drug-combination vs. pre-drug-combination change in VCPD between Visits 1 and 2 will be correlated with the post-drug-combination minus pre-drug-combination change in the pain severity score obtained from the BPI (score between 0 and 40; Gjeilo et al., 2007) between Visits 1 and 2.
Correlation between change in pupil constriction velocity (PCV) and change in the Brief Pain Inventory (BPI) score | 10 days
  To assess whether inter-individual differences in the drug-induced change in light-evoked PCV (in mm/s; Connely et al., 2014) predicts pain relief, the post-drug-combination minus pre-drug-combination change in PCV between Visits 1 and 2 (mm/s) will be correlated with the post-drug-combination minus pre-drug-combination change in the pain severity score obtained from the BPI (score between 0 and 40; Gjeilo et al., 2007) between Visits 1 and 2.
Correlation between change in saccadic peak velocity (SPV) and change in the Stanford Sleepiness Scale (SSS) | 10 days
  To assess whether inter-individual differences in the drug-induced change in SPV predicts self-reported sleepiness, the post-drug-combination vs pre-drug combination change in SPV (m/s) between Visits 1 and 2 (expressed as percentage of change) will be correlated with the post-drug-combination minus pre-drug-combination change in self-reported sleepiness assessed using the Stanford Sleepiness Scale (SSS; score between 1 and 7) between Visits 1 and 2.
Correlation between change in performance of the 2-back working memory task (2-WM) and change in the PROMIS Neuro-QOL score for cognitive function | 10 days
  To assess whether inter-individual differences in the drug-induced change in performance of the 2-WM (expressed as the discrimination index d-prime; Haatveit et al., 2010) predicts self-reported cognitive dysfunction, the post-drug-combination minus pre-drug-combination change in performance between Visits 1 and 2 will be correlated with the post-drug-combination minus pre-drug-combination change in self-reported cognitive dysfunction assessed using the short-form cognitive function measurement of the PROMIS Neuro-QOL (Quality of Life in Neurological Disorders) between Visits 1 and 2 (standardized T score for "cognitive function", having a mean of 50 and a standard deviation of 10 in a reference population).

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gjeilo KH, Stenseth R, Wahba A, Lydersen S, Klepstad P. Validation of the brief pain inventory in patients six months after cardiac surgery. J Pain Symptom Manage. 2007 Dec;34(6):648-56. doi: 10.1016/j.jpainsymman.2007.01.010. Epub 2007 Jul 16. PMID 17629665
- [Background] Kaida K, Takahashi M, Akerstedt T, Nakata A, Otsuka Y, Haratani T, Fukasawa K. Validation of the Karolinska sleepiness scale against performance and EEG variables. Clin Neurophysiol. 2006 Jul;117(7):1574-81. doi: 10.1016/j.clinph.2006.03.011. Epub 2006 May 6. PMID 16679057
- [Background] Comerchero MD, Polich J. P3a and P3b from typical auditory and visual stimuli. Clin Neurophysiol. 1999 Jan;110(1):24-30. doi: 10.1016/s0168-5597(98)00033-1. PMID 10348317
- [Background] Cruccu G, Aminoff MJ, Curio G, Guerit JM, Kakigi R, Mauguiere F, Rossini PM, Treede RD, Garcia-Larrea L. Recommendations for the clinical use of somatosensory-evoked potentials. Clin Neurophysiol. 2008 Aug;119(8):1705-1719. doi: 10.1016/j.clinph.2008.03.016. Epub 2008 May 16. PMID 18486546
- [Background] Askew RL, Cook KF, Keefe FJ, Nowinski CJ, Cella D, Revicki DA, Morgan DeWitt EM, Michaud K, Trence DL, Amtmann D. A PROMIS Measure of Neuropathic Pain Quality. Value Health. 2016 Jul-Aug;19(5):623-30. doi: 10.1016/j.jval.2016.02.009. Epub 2016 Apr 6. PMID 27565279
- [Background] Charier DJ, Zantour D, Pichot V, Chouchou F, Barthelemy JM, Roche F, Molliex SB. Assessing Pain Using the Variation Coefficient of Pupillary Diameter. J Pain. 2017 Nov;18(11):1346-1353. doi: 10.1016/j.jpain.2017.06.006. Epub 2017 Jul 13. PMID 28711635
- [Background] Connelly MA, Brown JT, Kearns GL, Anderson RA, St Peter SD, Neville KA. Pupillometry: a non-invasive technique for pain assessment in paediatric patients. Arch Dis Child. 2014 Dec;99(12):1125-31. doi: 10.1136/archdischild-2014-306286. Epub 2014 Sep 3. PMID 25187497
- [Background] Haatveit BC, Sundet K, Hugdahl K, Ueland T, Melle I, Andreassen OA. The validity of d prime as a working memory index: results from the "Bergen n-back task". J Clin Exp Neuropsychol. 2010 Oct;32(8):871-80. doi: 10.1080/13803391003596421. Epub 2010 Apr 9. PMID 20383801